CLINICAL TRIAL: NCT01115699
Title: Pilot Study of Repetitive Transcranial Magnetic Stimulation (rTMS) as Adjuvant Treatment in Patients With Non-remitting Depression: Third Stage of Citalopram/Escitalopram Study
Brief Title: Study of Repetitive Transcranial Magnetic Stimulation (rTMS) as Adjuvant Treatment for Depression
Acronym: rTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to funding constraints and recruitment was slower than was expected
Sponsor: Mayo Clinic (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Principal Investigator, David Mrazek, David Mrazek, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-000401
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Depression
Keywords: Depression; rTMS
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Repetitive Transcranial Magnetic Stimulation (Experimental): All subjects will receive 10 Hz repetitive transcranial magnetic stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (L-DLPFC) for a fixed-flexible period of 5 treatments per week for up to 6 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Active 10 Hz rTMS will be applied to the left dorsolateral prefrontal cortex (L-DLPFC) with an intensity of 120% motor threshold. The L-DLPFC location is defined as that area 5 cm anterior to the motor cortex for activation of abductor pollicis brevis. Subjects will receive a total of 3000 stimuli per session. The TMS trains are 4 seconds on and 26 seconds off for a total of 37 1/2 minutes. Treatment will occur 5 days per week for up to six weeks. Subjects will be monitored during rTMS for any side effects or adverse events.

SUMMARY:
The study will systematically investigate the use of repetitive transcranial magnetic stimulation (rTMS) in non-remitters of a selective serotonin reuptake inhibitor (SSRI) followed by a serotonin-norepinephrine reuptake inhibitor (SNRI) trial with the capacity to identify gene variants that predict rTMS response.

DETAILED DESCRIPTION:
This is the first study of its kind to systematically investigate the use of repetitive transcranial magnetic stimulation (rTMS) in non-remitters of a selective serotonin-reuptake inhibitor (SSRI) followed by an serotonin-norepinephrine reuptake inhibitor (SNRI) trial with the capacity to identify gene variants that predict rTMS response. The study is similar in design to the STAR*D study in that it will be the third treatment stage for a study of subjects with major depressive disorder (MDD). rTMS is a novel intervention which was FDA approved for treatment of MDD in October 2008 and was not clinically available at the time of the STAR*D study.

The primary aim of this pilot study is to provide 10 Hertz (Hz) repetitive transcranial magnetic stimulation (rTMS) applied to the left dorsolateral prefrontal cortex (L-DLPFC) as adjuvant treatment for depression in individuals who have not had a remission of their depressive symptoms after an 8 week trial of an SSRI (citalopram or escitalopram) followed by an 8 week trial of an SNRI, duloxetine and identify gene variants associated with improvement of their depressive symptoms.

ELIGIBILITY:
Inclusion Criteria

* Subjects whose depressive symptoms have not remitted during their participation in the "Pharmacokinetics and Pharmacodynamics of Citalopram and Escitalopram" study or the "Pharmacokinetics and Pharmacodynamics of Duloxetine" study
* Must be able to continue to take same dose of duloxetine through the course of the study

Exclusion Criteria

* A history of failure for respond to Electroconvulsive Therapy (ECT)
* Any metal in the head (except in mouth)
* Implanted medication pump or cardiac pacemaker
* Have had prior brain surgery
* Have unprovoked seizure disorder or family history of treatment resistant epilepsy
* Pregnancy
* Psychiatric hospitalization within the past two weeks
* Suicide attempt with hospitalization within past three months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mrazek, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repetitive Transcranial Magnetic Stimulation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Repetitive Transcranial Magnetic Stimulation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale for Depression (HRS-D17)
Description: The HRS-D17 questionnaire has 17 items. Each item on the questionnaire is scored on a 3 or 5 point scale, depending on the item. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression.
Time Frame: baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, and 6 weeks
Population: This study was stopped early due to funding constraints and recruitment was slower than was expected.
Arm/Group | Repetitive Transcranial Magnetic Stimulation
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Quick Inventory of Depressive Symptoms - Clinician Rating 16 Item (QIDS-C16)
Description: The QIDS-C16 measures 16 factors across 9 different criterion domains for major depression. Each of the four possible answers to each quiz is given an ascending numerical value from 0 to 3, and the total test score is the sum of the following:the highest number from questions 1-4 + the number from question 5 + the highest number from questions 6-9 + the total of each question from 10-14 + the highest number from questions 15-16.
  Screening test scoring ranges:
  * 0-5, No Depression Likely
  * 6-10, Possibly Mildly Depressed
  * 11-15, Moderate Depression
  * 16-20, Severe Depression
  * 21 or Over, Very Severe Depression
Time Frame: baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 5 weeks, and 6 weeks
Population: This study was stopped early due to funding constraints and recruitment was slower than was expected.
Arm/Group | Repetitive Transcranial Magnetic Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Repetitive Transcranial Magnetic Stimulation
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
This study was stopped early due to funding constraints and recruitment was slower than was expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No